CLINICAL TRIAL: NCT01492582
Title: Quadrivalent Human Papillomavirus (qHPV) Vaccine in Cancer Survivors: Cross Sectional Survey and Phase II Open-Label Vaccine Trial
Brief Title: Vaccine Therapy in Preventing Human Papillomavirus Infection in Younger Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Wendy Landier, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UAB-F141204009/UAB-X141204010; NCI-2011-03654 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1R01CA166559 (NIH); Merck-IISP#40083 (Other: Merck & Co.); COH-11034 (Other: City of Hope IRB)
Record Dates: First submitted 2011-12-12; First posted 2011-12-15 (Estimated); Results first posted 2020-04-30 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Cancer Survivor; Prevention of Human Papillomavirus Infection
MeSH Terms: interventions — Vaccines, Synthetic; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prevention (vaccine therapy) (Experimental): Patients receive quadrivalent human papillomavirus (types 6, 11, 16, and 18, for patients enrolled on or before 3/1/16) or nonavalent human papillomavirus (types 6, 11, 16, 18, 31, 33, 45, 52, and 58, for patients enrolled after 3/1/16) recombinant vaccine intramuscularly on day 1, at 8-12 weeks, and at 24-32 weeks.
  Interventions: Biological: quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine or nonavalent human papillomavirus vaccine (HPV 6, 11, 16, 18, 31, 33, 45, 52, 58); Other: laboratory biomarker analysis; Other: survey administration; Other: medical chart review

INTERVENTIONS:
Biological: quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine or nonavalent human papillomavirus vaccine (HPV 6, 11, 16, 18, 31, 33, 45, 52, 58) — Given IM
  Other Names: Gardasil; Gardasil 9
Other: laboratory biomarker analysis — Correlative studies
Other: survey administration — Ancillary studies
Other: medical chart review — Ancillary studies
  Other Names: chart review

SUMMARY:
This trial will comprehensively evaluate the human papillomavirus (HPV) vaccine in cancer survivors between 9 and 26 years of age by (1) determining the prevalence of HPV vaccine initiation among young cancer survivors, and (2) determining the immune response to and safety/tolerability of the quadrivalent and nonavalent HPV vaccine in young cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Using a cross-sectional survey approach, estimate the prevalence of HPV vaccine non-initiation: a) Examine sociodemographic, behavioral, and medical determinants of HPV vaccine non-initiation.

II. Using a single-arm, phase II, open-label, prospective longitudinal trial design, to evaluate the 3-dose HPV quadrivalent (HPV4) and nonavalent (HPV9) vaccine series and measure the following endpoints: a) Determine immunogenicity following the third and final vaccine dose; b) Identify clinical/host factors influencing immunogenicity; c) Determine the safety/tolerability of the HPV vaccine in cancer survivors.

III. Evaluate the persistence of antibody response at 2 years post vaccine initiation and identify clinical/host factors influencing response persistence.

OUTLINE:

AIM 1 (SURVEY): Patients (ages 18-26 years) or their parents (for patients ages 9-17 years) complete a survey regarding the patient's HPV vaccination status, knowledge of HPV-related disease, and factors important in making decisions regarding vaccination.

AIM 2 (VACCINE EVALUATION): Patients not previously immunized against HPV receive quadrivalent human papillomavirus recombinant vaccine (HPV-6, -11, -16, -18, for patients enrolled on or before 3/1/16) or the nonavalent human papillomavirus recombinant vaccine (HPV-6, -11, -16, -18, -31, -33, -45, -52, -58, for patients enrolled after 3/1/16) intramuscularly on day 1, at 8-12 weeks, and at 24-32 weeks.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1 (SURVEY) (AIM 1 is closed to enrollment)
* Cancer survivor
* Between 12 and 60 months after completion of cancer therapy (chemotherapy, radiation, hematopoietic cell transplant [HCT])
* Scheduled for a return clinic visit at one of the participating institutions
* English or Spanish-speaking
* Willing to provide informed consent/assent for study participation
* AIM 2 (VACCINE EVALUATION)
* Meets all inclusion criteria outlined in Aim 1
* Survey response indicated no prior history of HPV vaccination OR patient has no prior history of HPV vaccination by self - or parent/caregiver-report
* English or Spanish-speaking
* Medical clearance from treating clinician for study participation
* Agrees to return to participating institution for 3 HPV vaccine injections
* Willing to provide informed consent/assent for study participation

Exclusion Criteria:

* AIM 2 (VACCINE EVALUATION)
* Allergy to any component of the HPV vaccine including yeast and aluminum
* Thrombocytopenia (platelet count < 50K) or coagulation disorder that would contraindicate intramuscular injection
* Transfusion of blood products or intravenous immune globulin within 3 months of study entry
* Female, and a) currently pregnant or lactating, or b) of childbearing potential and unwilling to avoid pregnancy during the vaccine phase of study (beginning at Day 1 and continuing until at least 4 weeks after all 3 vaccine doses have been administered)

Ages: 9 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1499 (Actual)
Dates: Start 2012-07; Primary Completion 2019-02-08 (Actual); Study Completion 2020-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Landier, PhD, CRNP, Principal Investigator — University of Alabama at Birmingham
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope Medical Center, Duarte, California
  - Emory University School Of Medicine, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - Saint Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- [Derived] Landier W, Bhatia S, Wong FL, York JM, Flynn JS, Henneberg HM, Singh P, Adams K, Wasilewski-Masker K, Cherven B, Jasty-Rao R, Leonard M, Connelly JA, Armenian SH, Robison LL, Giuliano AR, Hudson MM, Klosky JL. Immunogenicity and safety of the human papillomavirus vaccine in young survivors of cancer in the USA: a single-arm, open-label, phase 2, non-inferiority trial. Lancet Child Adolesc Health. 2022 Jan;6(1):38-48. doi: 10.1016/S2352-4642(21)00278-9. Epub 2021 Nov 10. PMID 34767765
- [Derived] York JM, Klosky JL, Chen Y, Connelly JA, Wasilewski-Masker K, Giuliano AR, Robison LL, Wong FL, Hudson MM, Bhatia S, Landier W. Patient-Level Factors Associated With Lack of Health Care Provider Recommendation for the Human Papillomavirus Vaccine Among Young Cancer Survivors. J Clin Oncol. 2020 Sep 1;38(25):2892-2901. doi: 10.1200/JCO.19.02026. Epub 2020 Jun 18. PMID 32552278
- [Derived] Cherven B, Castellino SM, Chen Y, Wong FL, York JM, Wasilewski-Masker K, Hudson MM, Bhatia S, Klosky JL, Landier W. Intent and subsequent initiation of human papillomavirus vaccine among young cancer survivors. Cancer. 2019 Nov 1;125(21):3810-3817. doi: 10.1002/cncr.32379. Epub 2019 Jul 10. PMID 31291010
- [Derived] Klosky JL, Hudson MM, Chen Y, Connelly JA, Wasilewski-Masker K, Sun CL, Francisco L, Gustafson L, Russell KM, Sabbatini G, Flynn JS, York JM, Giuliano AR, Robison LL, Wong FL, Bhatia S, Landier W. Human Papillomavirus Vaccination Rates in Young Cancer Survivors. J Clin Oncol. 2017 Nov 1;35(31):3582-3590. doi: 10.1200/JCO.2017.74.1843. Epub 2017 Aug 24. PMID 28837404

RESULTS

PARTICIPANT FLOW:
Groups:
- Survey Arm: Patients (ages 18-26 years) or their parents (for patients ages 9-17 years) complete a survey regarding the patient's HPV vaccination status, knowledge of HPV-related disease, and factors important in making decisions regarding vaccination.
Period: Overall Study
Arm/Group | Prevention (Vaccine Therapy) | Survey Arm
Started (Type of vaccine based on standard of care at time of enrollment) | 453 (Consented to the vaccine arm (265 quadrivalent vaccine; 188 nonavalent vaccine)) | 1046 (Consented to the survey arm of the study)
Received First Quadrivalent Vaccine Dose | 254 | 0 (Does not apply)
Received First Nonavalent Vaccine Dose | 182 | 0
Completed | 384 (Received 3 vaccine doses and completed Month 7 blood draw (224 quadrivalent; 160 nonavalent)) | 982 (Returned evaluable survey)
Not Completed | 69 | 64

BASELINE CHARACTERISTICS:
Population: Participants who consented to the study.
Groups:
- Survey: Patients (ages 18-26 years) or their parents (for patients ages 9-17 years) complete a survey regarding the patient's HPV vaccination status, knowledge of HPV-related disease, and factors important in making decisions regarding vaccination.
- Total: Total of all reporting groups
Arm/Group | Prevention (Vaccine Therapy) | Survey | Total
Number analyzed (Participants) | 453 | 1046 | 1499
Age, Customized [Count of Participants; unit: Participants]
  9-15 years | 249 | 508 | 757
  16-26 years | 204 | 538 | 742
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 473 | 668
  Male | 258 | 573 | 831
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 142 | 194
  Not Hispanic or Latino | 400 | 900 | 1300
  Unknown or Not Reported | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 5 | 6
  Asian | 6 | 32 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Black or African American | 96 | 170 | 266
  White | 338 | 796 | 1134
  More than one race | 10 | 24 | 34
  Unknown or Not Reported | 2 | 16 | 18
Region of Enrollment [Number; unit: participants]
  United States | 453 | 1046 | 1499

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of HPV Vaccine Initiation in Cancer Survivors (Aim 1 [Survey])
Description: The prevalence of HPV vaccine initiation in cancer survivors ages 9 to 26 years
Time Frame: At baseline
Population: Participants who returned an evaluable survey
Measure: Count of Participants; unit: Participants
Groups:
- Survey Participants: Participants who consented to the survey aim of the study.
Arm/Group | Survey Participants
Number analyzed (Participants) | 982
Participants | 179

2. Primary Outcome: Immunogenicity of the HPV Vaccine in Cancer Survivors (Anti-HPV 16 and 18 Geometric Mean Titers) (Aim 2 [Vaccine Evaluation])
Description: To demonstrate the non-inferiority of the antibody responses to the HPV vaccine in cancer survivors ages 9 to 26 years when compared to antibody responses of age- and sex-matched historical healthy population.
Time Frame: 1 month following vaccination dose #3
Measure: Geometric Mean (Standard Deviation); unit: mMu/mL
Groups:
- Quadrivalent Anti-HPV 16, Male, Age 9-15 Years; Quadrivalent Anti-HPV 16, Female, Age 9-15 Years; Quadrivalent Anti-HPV 16, Male, Age 16-26 Years; Quadrivalent Anti-HPV 16, Female, Age 16-26 Years; Quadrivalent Anti-HPV 18, Male, Age 9-15 Years; Quadrivalent Anti-HPV 18, Female, Age 9-15 Years; Quadrivalent Anti-HPV 18, Male, Age 16-26 Years; Quadrivalent Anti-HPV 18, Female, Age 16-26 Years: Patients receive quadrivalent human papillomavirus (types 6, 11, 16, and 18, for patients enrolled on or before 3/1/16) recombinant vaccine intramuscularly on day 1, at 8-12 weeks, and at 24-32 weeks.
- Nonavalent Anti-HPV 16, Male, Age 9-15 Years; Nonavalent Anti-HPV 16, Female, Age 9-15 Years; Nonavalent Anti-HPV 16, Male, Age 16-26 Years; Nonavalent Anti-HPV 16, Female, Age 16-26 Years; Nonavalent Anti-HPV 18, Male, Age 9-15 Years; Nonavalent Anti-HPV 18, Female, Age 9-15 Years; Nonavalent Anti-HPV 18, Male, Age 16-26 Years; Nonavalent Anti-HPV 18, Female, Age 16-26 Years: Patients receive nonavalent human papillomavirus (types 6, 11, 16, 18, 31, 33, 45, 52, and 58, for patients enrolled after 3/1/16) recombinant vaccine intramuscularly on day 1, at 8-12 weeks, and at 24-32 weeks.
Arm/Group | Quadrivalent Anti-HPV 16, Male, Age 9-15 Years | Quadrivalent Anti-HPV 16, Female, Age 9-15 Years | Quadrivalent Anti-HPV 16, Male, Age 16-26 Years | Quadrivalent Anti-HPV 16, Female, Age 16-26 Years | Nonavalent Anti-HPV 16, Male, Age 9-15 Years | Nonavalent Anti-HPV 16, Female, Age 9-15 Years | Nonavalent Anti-HPV 16, Male, Age 16-26 Years | Nonavalent Anti-HPV 16, Female, Age 16-26 Years | Quadrivalent Anti-HPV 18, Male, Age 9-15 Years | Quadrivalent Anti-HPV 18, Female, Age 9-15 Years | Quadrivalent Anti-HPV 18, Male, Age 16-26 Years | Quadrivalent Anti-HPV 18, Female, Age 16-26 Years | Nonavalent Anti-HPV 18, Male, Age 9-15 Years | Nonavalent Anti-HPV 18, Female, Age 9-15 Years | Nonavalent Anti-HPV 18, Male, Age 16-26 Years | Nonavalent Anti-HPV 18, Female, Age 16-26 Years
Number analyzed (Participants) | 65 | 51 | 65 | 28 | 53 | 41 | 32 | 23 | 66 | 54 | 68 | 30 | 50 | 41 | 32 | 28
mMu/mL | 16134.57 (14722.06) | 15209.73 (15638.30) | 8740.02 (9625.61) | 6107.32 (6609.07) | 16419.64 (14756.37) | 11763.60 (8082.14) | 10770.38 (11166.73) | 11522.87 (10443.38) | 3472.21 (3769.68) | 2638.33 (2695.70) | 1920.01 (2553.81) | 1009.90 (990.48) | 5599.80 (4522.19) | 3457.20 (2510.32) | 3013.39 (3194.84) | 3483.29 (6869.27)
Statistical Analysis 1: Comparison: Quadrivalent Anti-HPV 16, Male, Age 9-15 Years; Historical Healthy Population Reference: QUADRIVALENT Male and female, all age groups: Merck Pub 9883616 (Gardasil Package Insert, April 2011, pp 24-26); Test type: Non-Inferiority — Non-inferiority required that the lower bound of the one-sided 99.688% confidence interval (CI) of the geometric mean titer (GMT) ratio was >0.5; lower bound one-sided CI of GMT ratio = 1.74 — GMT ratio = GMT (cancer survivor) / GMT (historical healthy population)
Statistical Analysis 2: Comparison: Quadrivalent Anti-HPV 16, Female, Age 9-15 Years; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; lower bound one-sided CI of GMT ratio = 1.76; GMT ratio = GMT (cancer survivor) / GMT (historical healthy population)
Statistical Analysis 3: Comparison: Quadrivalent Anti-HPV 16, Male, Age 16-26 Years; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; lower bound one-sided CI of GMT ratio = 2.15; GMT ratio = GMT (cancer survivor) / GMT (historical healthy population)
Statistical Analysis 4: Comparison: Quadrivalent Anti-HPV 16, Female, Age 16-26 Years; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; lower bound one-sided CI of GMT ratio = 1.00; GMT ratio = GMT (cancer survivor) / GMT (historical healthy population)
Statistical Analysis 5: Comparison: Quadrivalent Anti-HPV 18, Male, Age 9-15 Years; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; lower bound one-sided CI of GMT ratio = 1.52; GMT ratio = GMT (cancer survivor) / GMT (historical healthy population)
Statistical Analysis 6: Comparison: Quadrivalent Anti-HPV 18, Female, Age 9-15 Years; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; lower bound one-sided CI of GMT ratio = 1.48; GMT ratio = GMT (cancer survivor) / GMT (historical healthy population)
Statistical Analysis 7: Comparison: Quadrivalent Anti-HPV 18, Male, Age 16-26 Years; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; lower bound one-sided CI of GMT ratio = 2.48; GMT ratio = GMT (cancer survivor) / GMT (historical healthy population)
Statistical Analysis 8: Comparison: Quadrivalent Anti-HPV 18, Female, Age 16-26 Years; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; lower bound one-sided CI of GMT ratio = 1.00; GMT ratio = GMT (cancer survivor) / GMT (historical healthy population)
Statistical Analysis 9: Comparison: Nonavalent Anti-HPV 16, Male, Age 9-15 Years; Historical Healthy Population Reference: NONAVALENT Girls 9-15, Boys 9-15, Women 16-26: Petersen LK, Restrepo J, Moreira ED, Jr., et al. Impact of baseline covariates on the immunogenicity of the 9-valent HPV vaccine - A combined analysis of five phase III clinical trials. Papillomavirus Res. 2017;3:105-115;; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; lower bound one-sided CI GMT ratio = 1.23; GMT ratio = GMT (cancer survivor) / GMT (historical healthy population)
Statistical Analysis 10: Comparison: Nonavalent Anti-HPV 16, Female, Age 9-15 Years; [analysis description as in outcome 2, analysis 9]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; lower bound one-sided CI of GMT ratio = 1.12; GMT ratio = GMT (cancer survivor) / GMT (historical healthy population)
Statistical Analysis 11: Comparison: Nonavalent Anti-HPV 16, Male, Age 16-26 Years; Historical Healthy Population Reference: NONAVALENT Men 16-26: Castellsague X, Giuliano AR, Goldstone S, et al. Immunogenicity and safety of the 9-valent HPV vaccine in men. Vaccine. 2015;33(48):6892-6901. (HM data); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; lower bound one-sided CI of GMT ratio = 1.46; GMT ratio = GMT (cancer survivor) / GMT (historical healthy population)
Statistical Analysis 12: Comparison: Nonavalent Anti-HPV 16, Female, Age 16-26 Years; [analysis description as in outcome 2, analysis 9]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; lower bound one-sided CI of GMT ratio = 1.61; GMT ratio = GMT (cancer survivor) / GMT (historical healthy population)
Statistical Analysis 13: Comparison: Nonavalent Anti-HPV 18, Male, Age 9-15 Years; [analysis description as in outcome 2, analysis 9]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; lower bound one-sided CI of GMT ratio = 1.39; GMT ratio = GMT (cancer survivor) / GMT (historical healthy population)
Statistical Analysis 14: Comparison: Nonavalent Anti-HPV 18, Female, Age 9-15 Years; [analysis description as in outcome 2, analysis 9]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; lower bound one-sided CI of GMT ratio = 1.10; GMT ratio = GMT (cancer survivor) / GMT (historical healthy population)
Statistical Analysis 15: Comparison: Nonavalent Anti-HPV 18, Male, Age 16-26 Years; [analysis description as in outcome 2, analysis 11]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; lower bound one-sided CI of GMT ratio = 1.65; GMT ratio = GMT (cancer survivor) / GMT (historical healthy population)
Statistical Analysis 16: Comparison: Nonavalent Anti-HPV 18, Female, Age 16-26 Years; [analysis description as in outcome 2, analysis 9]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; lower bound one-sided CI of GMT ratio = -0.44; GMT ratio = GMT (cancer survivor) / GMT (historical healthy population)

3. Primary Outcome: Safety/Tolerability of the HPV Vaccine in Cancer Survivors (Aim 2 [Vaccine Evaluation])
Description: To demonstrate comparable safety/tolerability of the HPV vaccine in cancer survivors ages 9 to 26 years when compared to age- and sex-matched general population.
Time Frame: Dose 1 through Month 7
Population: Note: 254 participants received the first dose of the quadrivalent vaccine. However, one participant never returned to clinic or returned phone calls after receiving the first vaccine. No follow-up information is available for this participant so only 253 participants are reported in this group.
Measure: Number; unit: participants
Groups:
- Prevention (Vaccine Therapy)- Quadrivalent: Patients receive quadrivalent human papillomavirus (types 6, 11, 16, and 18, for patients enrolled on or before 3/1/16) recombinant vaccine intramuscularly on day 1, at 8-12 weeks, and at 24-32 weeks.
- Nonavalent Vaccine: Patients receive nonavalent human papillomavirus (types 6, 11, 16, 18, 31, 33, 45, 52, and 58, for patients enrolled after 3/1/16) recombinant vaccine intramuscularly on day 1, at 8-12 weeks, and at 24-32 weeks.
Arm/Group | Prevention (Vaccine Therapy)- Quadrivalent | Nonavalent Vaccine
Number analyzed (Participants) | 253 | 182
participants
  Injection site - Pain, any | 90 | 84
  Injection site - Swelling, any | 15 | 15
  Injection site - Erythema, any | 15 | 17
  Systemic - Headache | 51 | 33
  Systemic - Fever | 17 | 15
  Systemic - Nausea | 29 | 41
  Systemic - Dizziness | 5 | 2
  Systemic - Fatigue | 47 | 24
Statistical Analysis 1: Comparison: Prevention (Vaccine Therapy)- Quadrivalent; Injection site - Pain, any; Injection site - Swelling, any; Injection site - Erythema, any; Systemic - Nausea Historical Healthy Population: Reported from Gardasil Package Insert 04/2015, Tables 1, 2, 5, and 6; Test type: Superiority; p < 0.001, Chi-squared, Corrected
Statistical Analysis 2: Comparison: Prevention (Vaccine Therapy)- Quadrivalent; Systemic - Fever Historical Healthy Population: Reported from Gardasil Package Insert 04/2015, Tables 1, 2, 5, and 6; Test type: Superiority; p = 0.03, Chi-squared, Corrected
Statistical Analysis 3: Comparison: Prevention (Vaccine Therapy)- Quadrivalent; Systemic - Dizziness Historical Healthy Population: Reported from Gardasil Package Insert 04/2015, Tables 1, 2, 5, and 6; Test type: Superiority; p = 0.48, Chi-squared, Corrected
Statistical Analysis 4: Comparison: Nonavalent Vaccine; Injection site - Pain, any; Injection site - Swelling, any; Injection site - Erythema, any; Systemic - Nausea; Systemic - Fatigue Historical Healthy Population - As reported by Moreira et. al, 2016, Pediatrics, Table 5; Test type: Superiority; p < 0.001, Chi-squared, Corrected
Statistical Analysis 5: Comparison: Nonavalent Vaccine; Systemic - Headache Historical Healthy Population - As reported by Moreira et. al, 2016, Pediatrics, Table 5; Test type: Superiority; p = 0.07, Chi-squared, Corrected
Statistical Analysis 6: Comparison: Nonavalent Vaccine; Systemic - Fever Historical Healthy Population - As reported by Moreira et. al, 2016, Pediatrics, Table 5; Test type: Superiority; p = 0.28, Chi-squared, Corrected
Statistical Analysis 7: Comparison: Nonavalent Vaccine; Systemic - Dizziness Historical Healthy Population - As reported by Moreira et. al, 2016, Pediatrics, Table 5; Test type: Superiority; p = 0.45, Fisher Exact

ADVERSE EVENTS:
Time Frame: Other (Not Including Serious) Adverse Events: Nonavalent: 7 days after each vaccine dose Quadrivalent: 14 days after each vaccine dose Serious Adverse Events were reported up to Month 7 (no SAEs occurred within 7-14 days of each vaccine dose).
Description: No adverse events are reported for the survey arm participants as adverse events were not monitored/assessed for participants in this arm.
  Note: 254 participants received the first dose of the quadrivalent vaccine. However, one participant never returned to clinic or returned phone calls after receiving the first vaccine. No follow-up information is available for this participant so only 253 participants are reported in this group.
Groups:
- Prevention (Vaccine Therapy)- Nonavalent Vaccine: Patients receive nonavalent human papillomavirus (types 6, 11, 16, 18, 31, 33, 45, 52, and 58, for patients enrolled after 3/1/16) recombinant vaccine intramuscularly on day 1, at 8-12 weeks, and at 24-32 weeks.
Arm/Group | Prevention (Vaccine Therapy)- Quadrivalent | Prevention (Vaccine Therapy)- Nonavalent Vaccine
All-Cause Mortality (participants affected / at risk) | 0/253 | 0/182
Serious Adverse Events (participants affected / at risk) | 11/253 | 7/182
Other Adverse Events (participants affected / at risk) | 129/253 | 108/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevention (Vaccine Therapy)- Quadrivalent (N=253) | Prevention (Vaccine Therapy)- Nonavalent Vaccine (N=182)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Relapse of primary cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Subsequent malignant neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1
Hospitalization for musculoskeletal issue (Musculoskeletal and connective tissue disorders) | 4 | 0
Hospitalization for endocrine disorder (Endocrine disorders) | 2 | 0
Hospitalization for fluid-electrolyte disorder (Metabolism and nutrition disorders) | 0 | 1
Hospitalization for neurologic disorder (Nervous system disorders) | 0 | 1
Hospitalization for psychiatric disorder (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prevention (Vaccine Therapy)- Quadrivalent (N=253) | Prevention (Vaccine Therapy)- Nonavalent Vaccine (N=182)
Injection Site Pain or Tenderness, any (General disorders) | 90 | 84
Injection Site Swelling, any (General disorders) | 15 | 15
Injection Site Erythema, any (General disorders) | 15 | 17
Headache (General disorders) | 51 | 33
Fever (≥100.0⁰F) (General disorders) | 17 | 15
Nausea (Gastrointestinal disorders) | 29 | 41
Fatigue (General disorders) | 47 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-03-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT01492582/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT01492582/ICF_001.pdf